CLINICAL TRIAL: NCT02341365
Title: Impact of Vitamin D Levels on Ovarian Reserve and Ovarian Response to Controlled Stimulation in Egg Donors
Brief Title: Vitamin D Influence on Oocyte Donation
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 1406-MAD-035-JG
Record Dates: First submitted 2014-11-07; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Disorder of Phosphate, Calcium and Vitamin D Metabolism; Female Infertility Due to Diminished Ovarian Reserve; Hormonal Requirement; Reproductive Disorder
Keywords: Egg donation; vitaminD; ovarian reserve; ovarian stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: vitamin D,AMH, AFC, reproductive outcome egg recipients — observational study of 269 donnors

SUMMARY:
Objective: To investigate the correlation between total and bioavailable serum 25-OH vitamin D, ovarian reserve and ovarian response to controlled stimulation in egg donors.

DETAILED DESCRIPTION:
Design: Retrospective study. Setting: University affiliated private IVF center. Intervention: Serum analysis of vitamin D, bioavailable vitamin D, antimullerian hormone (AMH), antral follicular count (AFC), reproductive outcome of oocytes recipients Main outcome measure: AMH, AFC, number of oocytes retrieved and number of mature oocytes, pregnancy and implantation rate of donated oocytes'recipients.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian race,
* between 18 and 34 years of age,
* all donors had normal menstrual cycles of 26-34 days,
* normal weight range (BMI 18- 25 Kg/m2),
* normal uterus and ovaries on transvaginal ultrasound (no signs of polycystic ovarian syndrome), and
* an antral follicle count (AFC) >10,
* normal karyotype

Exclusion Criteria:

* current or past exposure to radiation or hazardous chemical substances,
* history of drug use,
* family history of hereditary chromosomal diseases,
* sexually transmitted diseases

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: oocytes' donors who underwent ovarian stimulation cycles in our clinic from June 2013 to April 2014
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Numbers of oocytes retrieved | 2 months

SECONDARY OUTCOMES:
implantation rate | 2 months
pregnancy rate | 2 months
AFC | 2 months
number of mature oocytes | 2 months
AMH | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio García Velasco, Professor, Principal Investigator — IVI Madrid

REFERENCES:
- [Result] Holick MF et al. Endocrine Society. Evaluation, treatment, prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011;96:1911-1930 Rudick B et al. Characterizing the influence of vitamin D levels on IVF outcomes. Hum Reprod. 2012;27:3321-7 Polyzos NP et al. Vitamin D deficiency and pregnancy rates in women undergoing single embryo, blastocyst stage, transfer (SET) for IVF/ICSI. Hum Reprod. 2014;29:2032-40 Franasiak JM et al. Vitamin D levels do not affect IVF outcomes following the transfer of euploid blastocysts. Am J Obstet Gynecol 2014;211:x.ex-x.ex Fabris A, Pacheco A, Cruz M, Puente JM, Fatemi H, Garcia-Velasco JA. Impact of circulating levels of total and bioavailable serum vitamin D on pregnancy rate in egg donation recipients. Fertil Steril. 2014. Irani M, Merhi Z. Role of vitamin D in ovarian physiology and its implication in reproduction: a systematic review. Fertil Steril. 2014 ;102:460-468